CLINICAL TRIAL: NCT04545788
Title: A Randomized, Controlled, Multi-center Clinical Trial of Short Course Treatment for Newly Diagnosed Rifampicin Resistant Tuberculosis
Brief Title: Randomized Controlled Multi-center Short Course Treatment for Rifampicin Resistant Tuberculosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Chu naihu, TB Director, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCP-TB
Record Dates: First submitted 2020-08-31; First posted 2020-09-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, rifampin resistant, oral, shorter.
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Active Comparator): 4-6 INH EMB PZA Pto AM Cfz Mfx / 5 EMB PZA Cfz Mfx (INH: Isoniazid, EMB: Ethambutol, PZA: Pyrazinamide, Pto: Prothionamide, AM: Amikacin, Cfz: Clofazimine, Mfx: Moxifloxacin) A group is the control group which includes injectable drugs (AM).
  Interventions: Drug: Total oral short-term therapy that includes linezolid, bedaquiline and/or cycloserine.
- B (Experimental): 4-6 INH EMB PZA Pto LZD Cfz Mfx / 5 EMB PZA Cfz Mfx (INH: Isoniazid, EMB: Ethambutol, PZA: Pyrazinamide, Pto: Prothionamide, LZD: Linezolid, Cfz: Clofazimine, Mfx: Moxifloxacin) B group is the experimental groups which is total oral short-term therapy.
  Interventions: Drug: Total oral short-term therapy that includes linezolid, bedaquiline and/or cycloserine.
- C (Experimental): 4-6 BDQ LZD MFX CS CFZ / 5MFX CS CFZ (BDQ: Bedaquiline, LZD: Linezolid, Mfx: Moxifloxacin, CS: Cycloserine, Cfz: Clofazimine) C group is another experimental groups which is also total oral short-term therapy, and includes new anti-TB drugs: BDQ.
  Interventions: Drug: Total oral short-term therapy that includes linezolid, bedaquiline and/or cycloserine.

INTERVENTIONS:
Drug: Total oral short-term therapy that includes linezolid, bedaquiline and/or cycloserine. — AM is the traditional anti-TB drugs. Linezolid, bedaquiline and/or cycloserine, that might have potential efficacy of replacing injectable anti-TB drugs, are included into the total oral short-term therapy, and replace AM.

SUMMARY:
This study is a randomized, controlled, multi-center clinical study. The main purpose of this study was to study the efficacy and safety data of total oral short-term therapy as an alternative to injection in the treatment of newly diagnosed RR-TB patients.

DETAILED DESCRIPTION:
A group: 4-6 INH EMB PZA Pto AM Cfz Mfx / 5 EMB PZA Cfz Mfx B group: 4-6 INH EMB PZA Pto LZD Cfz Mfx / 5 EMB PZA Cfz Mfx C group: 4-6 BDQ LZD MFX CS CFZ / 5MFX CS CFZ (INH: Isoniazid, EMB: Ethambutol, PZA: Pyrazinamide, Pto: Prothionamide, AM: Amikacin, Cfz: Clofazimine, Mfx: Moxifloxacin, LZD: Linezolid, BDQ: Bedaquiline, CS: Cycloserine) A group is the control group which includes injectable drugs (AM). B group and C group are the experimental groups which are total oral short-term therapy.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent and accepted follow-up;
* the age is between 18 and 65 years old, both male and female, including inpatients and outpatients;
* no use of anti tuberculosis drugs, or use of anti tuberculosis drugs less than 1 month;
* the results of molecular biology test confirmed rifampicin resistance or MDR-TB patients;
* chest CT examination confirmed pulmonary tuberculosis, pulmonary lesions, or cavity;
* premenopausal women had negative pregnancy urine test and agreed to use high-efficiency contraceptive measures during the study period.

Exclusion Criteria:

* drug sensitivity test or molecular drug sensitivity results show that the drug resistance (except isoniazid) or any component of the drug has a history of allergy, or is taking any drug that is contraindicated to the drug in the short-term treatment program;
* severe renal insufficiency (creatinine clearance rate (CrCl) less than 30 ml / min).
* liver function impairment (ALT and / or AST level 3 times higher than the upper limit of laboratory reference value, if it is temporary increase, it can be included after treatment recovery);
* those who are unable to participate in or comply with the treatment and follow-up;
* Q-T interval > 450 millisecond;
* have a history of cardiovascular diseases or are suffering from such diseases as heart failure, hypertension (poor blood pressure control), arrhythmia or post myocardial infarction state;
* pregnant or lactating women;
* those who are unable to take oral drugs;
* those who are currently participating in other clinical trials;
* patients with HIV positive or active viral hepatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Culture of Mycobacterium tuberculosis in sputum. | Through study completion, an average of 1 year.
  Mycobacterium tuberculosis culture of sputum will be carried out every month to understand the negative conversion rate and time of sputum bacteria, and then to understand the cure rate of patients. The final aim is to understand the efficacy of the total oral short-term anti-tuberculosis regimen.

SECONDARY OUTCOMES:
Adverse effect. | Through study completion, an average of 1 year.
  All the types and frequency of adverse reactions that related to anti-tuberculosis drug were collected.

CONTACTS AND LOCATIONS:
Overall Officials: NAIHUI CHU, Doctor, Principal Investigator — Beijing Chest Hospital affiliated to Capital Medical University
Locations (1):
- Beijing Chest Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du Y, Qiu C, Chen X, Wang J, Jing W, Pan H, Chen W, Liu Y, Li C, Xi X, Yin H, Zeng J, Zhang X, Xu T, Wang Q, Guo R, Wang J, Pang Y, Chu N. Treatment Outcome of a Shorter Regimen Containing Clofazimine for Multidrug-resistant Tuberculosis: A Randomized Control Trial in China. Clin Infect Dis. 2020 Aug 14;71(4):1047-1054. doi: 10.1093/cid/ciz915. PMID 31549147
- [Background] Wang Q, Pang Y, Jing W, Liu Y, Wang N, Yin H, Zhang Q, Ye Z, Zhu M, Li F, Liu P, Wu T, Chen W, Wu W, Qin Z, Qiu C, Deng Q, Xu T, Wang J, Guo R, Du Y, Wang J, Huang H, Chen X, Chu N. Clofazimine for Treatment of Extensively Drug-Resistant Pulmonary Tuberculosis in China. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e02149-17. doi: 10.1128/AAC.02149-17. Print 2018 Apr. PMID 29378718
- [Background] Wang J, Pang Y, Jing W, Chen W, Guo R, Han X, Wu L, Yang G, Yang K, Chen C, Jiang L, Cai C, Dou Z, Diao L, Pan H, Wang J, Du F, Xu T, Wang L, Li R, Chu N. Efficacy and safety of cycloserine-containing regimens in the treatment of multidrug-resistant tuberculosis: a nationwide retrospective cohort study in China. Infect Drug Resist. 2019 Apr 3;12:763-770. doi: 10.2147/IDR.S194484. eCollection 2019. PMID 31040707
- [Background] Pang Y, Jing W, Lu J, Zong Z, Huo F, Dong L, Dai G, Li Y, Huang H, Chu N. No in vitro synergistic effect of bedaquiline combined with fluoroquinolones, linezolid, and clofazimine against extensively drug-resistant tuberculosis. Diagn Microbiol Infect Dis. 2019 Aug;94(4):361-364. doi: 10.1016/j.diagmicrobio.2019.02.012. Epub 2019 Feb 19. PMID 30876684